CLINICAL TRIAL: NCT01432158
Title: A Detailed Kinetics Study to Assess the Antibody and the B Cell Response to Either a 13-valent Conjugate Vaccine or a 23-valent Plain Pneumococcal Polysaccharide Vaccine Administered to Healthy Adults Without Prior Pneumococcal Vaccination
Brief Title: Pneumococcal Adult Kinetics Study - Understanding the B Cell Response to Pneumococcal Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mason Medical Research Trust (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011/04B
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Pneumococcal Disease
Keywords: Invasive pneumococcal disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCV-13 group (Experimental): 1 dose of Prevenar-13
  Interventions: Biological: Prevenar 13
- PPV-23 group (Experimental): 1 dose of Pneumovax-II
  Interventions: Biological: Pneumovax II

INTERVENTIONS:
Biological: Prevenar 13 — This vaccine will be given to healthy adults without prior pneumococcal vaccination.
  Arms: PCV-13 group
Biological: Pneumovax II — This vaccine will be given to healthy adults without prior pneumococcal vaccination.
  Arms: PPV-23 group

SUMMARY:
This is an open-label phase III clinical trial. The purpose of this trial is to investigate in detail the kinetics of the immune response to Prevenar-13, a pneumococcal conjugate vaccine, compared to Pneumovax-II, a pneumococcal plain polysaccharide vaccine. With their consent, healthy adults (n=2 in each group) aged over 18 years who have not received any pneumococcal vaccine in the past will receive either vaccine at their first visit. Blood will be taken before vaccination and at day 0,1,2,4,6,8,10,12,14,16,18,20,23,26,30,35 as well as 2,6 and 12 months following vaccination. With specific consent, a small volume of blood will be used to store DNA and RNA for analysis of the genetic associations with immune responses and adverse reactions to vaccines as well as the RNA expression following a vaccination. Serum or plasma will be used to assess antibody level and available whole blood will be used for B cell assays and to examine immunoglobulin gene usage in B cells.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age.
* Participant is willing and able to give informed consent for participation after the nature of the study has been explained;
* In good health as determined by:

  * medical history
  * history-directed physical examination
  * clinical judgment of the investigator
* Able (in the Investigators opinion) and willing to comply with all study requirements including be available for all the visits scheduled in the study
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Have previously received a pneumococcal vaccine
* Have received vaccination with a vaccine containing either CRM197 or diphtheria toxoid within the past 12 months,
* Have had previous ascertained disease caused by C. diphtheriae, or S. pneumoniae in the past 5 years documented in their medical notes
* Have a history of any anaphylactic shock, asthma, urticaria or other allergic reaction after previous vaccinations or known hypersensitivity to any vaccine component;
* Have a known or suspected autoimmune disease or impairment /alteration of immune function resulting from (for example):

  * Receipt of immunostimulants
  * Congenital or acquired immunodeficiency, or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months or long-term systemic corticosteroid therapy (prednisolone or equivalent for more than two consecutive weeks within the past 3 months).
* Have a suspected or known HIV infection or HIV related disease;
* Have received blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 3 months
* Have a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time;
* Have any condition, which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.
* Participation in another clinical trial investigating a vaccine, a drug, a medical device, or a medical procedure
* Pregnancy as confirmed by a positive pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Frequency of serotype-specific B cell subsets determined by FACS. | within first month after vaccination
  To assess and compare the kinetics of serotype-specific B cell subsets following a dose of PCV-13 or PPCV-23 given to healthy adults.

SECONDARY OUTCOMES:
Pneumococcal serotype-specific geometric mean concentrations (GMC) | within first month after vaccination
  To assess and compare the kinetics of serotype-specific antibody (subclass) geometric mean concentrations (GMC) in response to a dose of PCV-13 or PPCV-23 given to healthy adults.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Pollard, BSc MBBS PhD MRCP FRCPCH, Principal Investigator — Department of Paediatrics, Oxford University
Locations (1):
- Oxford Vaccine Group, Oxford, United Kingdom